CLINICAL TRIAL: NCT05835453
Title: PATIENT SATISFACTION WITH AT-HOME DENTAL BLEACHING USING VIVERA OR ESSIX RETAINERS: A RANDOMIZED CLINICAL TRIAL
Brief Title: At-home Bleaching Using Clear Retainers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Collaborators: Align Technology, Inc. (Industry)
Responsible Party: Principal Investigator, Isabel Giráldez de Luis, Assistant Professor, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: URJC_IDIBO_1
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Tooth Discoloration; Tooth Sensitivity; Gingivitis; Satisfaction, Patient
Keywords: At-home tooth bleaching; Clear aligner; Tooth sensitivity; Gingival irritation; Patient´s satisfaction
MeSH Terms: conditions — Tooth Discoloration; Dentin Sensitivity; Gingivitis; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: This is a randomized, single blind (evaluators), split mouth and equivalence study.
Who Masked: Investigator, Outcomes Assessor
Masking Description: It will be a single-blind study in which only the evaluator will not know the designation of the groups because he has not participated in the study's randomization and implementation process. Due to the tray test and demonstration of the bleaching procedure, the operator and the participant cannot be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Essix-type retairner (Active Comparator): Two simple randomizations will be performed using a software program freely available online (www.sealedenvelop.com). For the first randomization, for each participant, the group (type of tray) will be randomized and it will always be applied to the participant's right hemiarch (n=40) according to the model: essix-type retairner or Vivera retainer. Subsequently, the second randomization will be carried out, which will define the alternate days for the use of essix-type retairner and Vivera retainer: Monday, Wednesday and Friday or Tuesday, Thursday and Saturday.
  Interventions: Other: Whitening
- Vivera retainer (Active Comparator): The patients will use the clear aligner on their right hemiarch and according to the second randomization it will be applied on Monday, Wednesday and Friday or Tuesday, Thursday and Saturday.
  Interventions: Other: Whitening

INTERVENTIONS:
Other: Whitening — Two syringes of 10% carbamide peroxide bleaching gel will be provided for use with each type of tray. Volunteers will be instructed to use the whitening gel once a day for 2 hours, for 3 days per week with each retainer, completing a total of 4 weeks of whitening procedure.

SUMMARY:
The aim of this project is to clinically evaluate patient satisfaction, whitening efficacy, tooth sensitivity, and gingival irritation during at-home whitening with 10% carbamide peroxide using an Essix-type retainer or a Vivera retainer.

DETAILED DESCRIPTION:
Forty patients (n=40) will be randomized as to which side will receive the type of bleaching tray, essix-type retairner or Vivera retainer. The at-home bleaching will be performed with 10% carbamide peroxide (Opalescence PF 10%) for 2 hours The treatment lasted 4 weeks, although as each retainer was worn every other day, the actual application time was 2 weeks. Patient´s satisfaction will be evaluated at baseline, after one, two weeks, and 4 weeks with an apropriate questionnaire using a visual analog scale (EVA 0-10). The color will be assessed at baseline, after one, two and four weeks using subjective color guides (VITA Classical and VITA Bleachguide 3D-MASTER) and a objective digital spectrophotometer (VITA Easyshade). The intensity and absolute risk of tooth sensitivity and gingival irritation will also be determined with a visual analog scale (EVA 0-10). Color change between groups will be compared by paired Student´s t-test. The absolute risk of tooth sensitivity and gingival irritation for both groups will be compared by McNemar test. Also, odds ratios, confidence intervals, and Spearman correlation will be determined. The intensity of tooth sensitivity, gingival irritation and patient´s satisfaction will be compared by paired Student´s t-test. The level of statistical significance accepted will be 5% for all analyses.

ELIGIBILITY:
The inclusion criteria will be the following:

* Patients over 18 years of age.
* Patients with vital teeth without restorations, single crowns, implants and/or bridges at the level of the anterior teeth.
* Absence of cavities in the teeth to be whitened.
* Patients with satisfactory oral hygiene, and periodontally healthy, who are not undergoing periodontal maintenance and who do not use chlorhexidine rinses. Patients with recessions without sensitivity are included.
* Absence of sensitivity, measured based on stimulation with the air from the syringe.
* Patients who are at least in A2-A3 color (Vita Classic Guide)

The exclusion criteria will be the following:

* Patients who have previously undergone whitening (less than 5 years).
* Patients undergoing orthodontic treatment.
* Patients with white spot or developmental alterations (dentinogenesis imperfecta, amelogenesis imperfecta) or with stains (tetracyclines or fluorosis).
* Patients with a history of trauma to anterior teeth.
* Patients who require internal whitening.
* Smokers.
* Pregnant or lactating women.
* Allergy to any component of whitening.
* Alterations of the oral mucosa (desquamative gingivitis, OLP, leukoplakias, etc.).
* Medical conditions considered by the researchers that may compromise the study or the individual safety of the patient.
* Patients with poor oral hygiene.
* Patients with previous hypersensitivity.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-14 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Patient´s satisfaction | Baseline, after one, two and four weeks
  It will be measured with a questionnaire using a visual analog scale (EVA), when a essix-type retairner or Vivera retainer is used to perform a at home bleaching treatment with 10% carbamide peroxide.

SECONDARY OUTCOMES:
Color change evaluation | Baseline, after one, two and four weeks
  The color will be assesed using subjetive color guides (VITA Classical and VITA 3D-MASTER) and a objetive digital spectrophotometer (VITA Easyshade).
Intensity and absolute risk of tooth sensitivity | Baseline, after one, two, four weeks, and at 1 month after bleaching treatment
  They will be determined by means of a visual analog scale (EVA), using a essix-type retairner or Vivera retainer, during at home bleaching treatment with 10% carbamide peroxide.
Intensity and absolute risk of gingival irritation | Baseline, after one, two, four weeks, and at 1 month after bleaching treatment
  They will be determined by means of a visual analog scale (EVA), using a essix-type retairner or Vivera retainer, during at home bleaching treatment with 10% carbamide peroxide.

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Dental Iturralde, Tafalla, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Almeida LC, Riehl H, Santos PH, Sundfeld ML, Briso AL. Clinical evaluation of the effectiveness of different bleaching therapies in vital teeth. Int J Periodontics Restorative Dent. 2012 Jun;32(3):303-9. PMID 22408775
- [Background] Carneiro TS, Favoreto MW, Bernardi LG, Sutil E, Wendlinger M, Centenaro GG, Reis A, Loguercio AD. Gingival irritation in patients submitted to at-home bleaching with different cutouts of the bleaching tray: a randomized, single-blind clinical trial. Clin Oral Investig. 2022 Jun;26(6):4381-4390. doi: 10.1007/s00784-022-04401-4. Epub 2022 Feb 7. PMID 35128627